CLINICAL TRIAL: NCT03957564
Title: Liquid Biopsy in Monitoring the Neoadjuvant Chemotherapy and Operation in Patients With Resectable or Locally Advanced Gastric or Gastro-oesophageal Junction Cancer
Brief Title: Liquid Biopsy in Monitoring the Neoadjuvant Chemotherapy and Operation in Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Qinghai University (Other)
Responsible Party: Principal Investigator, Jiuda Zhao, Professor, Affiliated Hospital of Qinghai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHQU-2019002
Record Dates: First submitted 2019-05-07; First posted 2019-05-21 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Gastric Cancer; Gastro-oesophageal Junction Cancer
Keywords: Gastric cancer; Gastro-oesophageal junction cancer; Neoadjuvant chemotherapy; Radical gastrectomy; Circulating tumor cells; Circulating tumor DNA; Circulating cell free DNA
MeSH Terms: conditions — Stomach Neoplasms; Neoplastic Cells, Circulating | interventions — Neoadjuvant Therapy; Circulating Tumor DNA; Cell-Free Nucleic Acids; CA-19-9 Antigen; CA-72-4 antigen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients receiving neoadjuvant chemotherapy. (Experimental): 1. Compare the monitoring of CTC, ctDNA and cfDNA with the results of CT scan and the blood level of CEA ,CA19-9 and CA72-4 tumor markers to explore the clinical value of dynamic detection of CTC, ctDNA and cfDNA in neoadjuvant chemotherapy and operation for locally advanced or resectable gastric or gastro-oesophageal junction cancer.
  2. Explore the clinical value of different types of CTC in neoadjuvant chemotherapy and Operation for locally advanced or resectable gastric or gastro-oesophageal junction cancer. CTC can be classified into three types: epithelial CTC, mesenchymal CTC, hybrids CTC.
  3. Explore the consistency between plasma ctDNA and tumor related DNA in pathological tissues after operation.
  4. To explore the relationship between the dynamic changes of plasma CTC, ctDNA and cfDNA levels and the prognosis of patients after operation.
  Interventions: Drug: Neoadjuvant chemotherapy with PSOX regimen.; Other: Detect the imaging data and levels of CTC, ctDNA, cfDNA, CEA, CA19-9, CA72-4 in plasma.; Other: Detect the tumor related DNA in pathological tissues after operation.; Other: Follow-up of DFS and OS in patients with gastric cancer after operation.

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy with PSOX regimen. — Resectable gastric or gastro-oesophageal junction cancer patients receiving neoadjuvant chemotherapy with PSOX（Paclitaxel+Oxaliplatin+S1）regimen.
  The details are as follows:
  Paclitaxel 135mg/m2 d1, Oxaliplatin 85mg/m2 d1, S1 40-60mg/m2 twice daily, d1-14 , 21 days is one cycle.
Other: Detect the imaging data and levels of CTC, ctDNA, cfDNA, CEA, CA19-9, CA72-4 in plasma. — Detect the imaging data and levels of CTC, ctDNA, cfDNA, CEA, CA19-9, CA72-4 in 3 time points：Before neoadjuvant chemotherapy, After 2-3 cycles of neoadjuvant chemotherapy, 10 days after operation.
Other: Detect the tumor related DNA in pathological tissues after operation. — Detect the tumor related DNA in pathological tissues after operation.
Other: Follow-up of DFS and OS in patients with gastric cancer after operation. — Follow-up of DFS and OS in patients with locally advanced or resectable gastric or gastro-oesophageal Junction cancer.

SUMMARY:
To explore the clinical value of dynamic detection of circulating tumor cells(CTCs), circulating tumor DNA(ctDNA) and cell-free DNA(cfDNA) in neoadjuvant chemotherapy and operation of resectable or locally advanced gastric or gastro-oesophageal junction cancer.

DETAILED DESCRIPTION:
Gastric cancer(GC) is one of the common malignant tumors in world, with relatively high incident rate and mortality among the population. Neoadjuvant chemotherapy is often needed before operation for locally advanced or resectable gastric or gastro-oesophageal junction cancer. Neoadjuvant chemotherapy should be combined with platinum and fluorouracil, or paclitaxel should be added on the basis of platinum and fluorouracil. The efficacy of neoadjuvant chemotherapy for GC patients is usually evaluated by computer tomography(CT) scans with RECIST 1.1 criteria and the blood level of carcinoembryonic antigen(CEA),CA19-9 (carbohydrate antigen 19-9)and CA72-4(carbohydrate antigen 72-4) tumor markers.

CTC originating from solid tumors are related to hematogenous metastatic spread to distant sites. Therefore, CTC analysis has clinical relevance as a biomarker to noninvasively monitor cancer progression and guide therapy.Moreover, ctDNA is a part of cfDNA derived from apoptotic, necrotic or secreted DNA fragments of tumor cells, ctDNA contains the same genetic defects as the tumor DNA of its origin, such as point mutation and rearrangement. We speculate CTC, ctDNA and cfDNA are new biomarkers for tumor, which can guide neoadjuvant chemotherapy and surgical treatment for patients with locally advanced or resectable gastric or gastro-oesophageal junction cancer.

In this study, investigators will compare the clinical value of the dynamic detection of CTC, ctDNA and cfDNA with CEA ,CA19-9 and CA72-4 tumor markers and CT scan according the RECIST 1.1 criteria in neoadjuvant chemotherapy and operation for resectable or locally advanced gastric or gastro-oesophageal junction cancer. Investigators will also explore the relationship between the dynamic changes of CTC, ctDNA and cfDNA and the prognosis of patients after operation. The results will provide lots of meaningful information which may further improve the treatment of locally advanced or resectable gastric or gastro-oesophageal junction cancer.

ELIGIBILITY:
Inclusion Criteria：

1. Patients with resectable or locally advanced gastric or gastro-oesophageal junction cancer(>T1 and N+) without distant metastases (M0).
2. Pathological examination confirmed gastric or gastro-oesophageal junction cancer (adenocarcinoma, signet ring cell carcinoma, mucinous adenocarcinoma, squamous cell carcinoma, regardless of the degree of tissue differentiation).
3. Ambulatory males or females, age ≥ 18 years.
4. Karnofsky Performance Score (KPS) ≥70 or ECOG(Eastern Cooperative Oncology Group) performance status: 0 or 1.
5. Patients who can tolerate PSOX neoadjuvant chemotherapy.
6. Planning to undergo radical gastrectomy after neoadjuvant chemotherapy.
7. With cancer lesions that can be measured according to RECIST 1.1 criteria.
8. No prior antitumor treatment is allowed, including chemotherapy, radiotherapy, immune therapy or target therapy.
9. Adequate organ function as defined below: Hemoglobin ≥ 9 g/dl, Absolute neutrophil count(ANC） ≥ 1.5×109/L, Platelets ≥ 100*109/L, Alkaline phosphatase( ALP) ≤ 2.5×ULN,Total bilirubin（TBIL）≤ 1.5×ULN(upper limit of normal), Renal Serum Creatinine < 1.5 ULN, Serum Albumin ≥ 30g/l.

Exclusion criteria:

1. Female in pregnancy or lactation, or refuse to receive contraception measures during chemotherapy.
2. With distant metastasis or peritoneal dissemination diagnosed by CT/EUS(endoscopic ultrasonography).
3. Underwent prior antitumor treatment, including chemotherapy, radiotherapy, immune therapy or target therapy.
4. Serious uncontrolled intercurrent infections or other serious uncontrolled concomitant disease or condition that would make the subject inappropriate for study participation.
5. Clinically serious cardiac disease or pulmonary dysfunction.
6. Refuse to provide blood/tissue sample.
7. Other situation to be judged not adaptive to the study by investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-28 (Actual); Primary Completion 2022-05-20 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
Numbers of CTC pre- and post- neoadjuvant chemotherapy and after operation. | 2 years
  Numbers of CTC pre- and post- neoadjuvant chemotherapy and after operation.
Types of CTC pre- and post- neoadjuvant chemotherapy and after operation. | 2 years
  Types of CTC pre- and post- neoadjuvant chemotherapy and after operation.
Mutation rate of ctDNA pre- and post- neoadjuvant chemotherapy and after operation. | 2 years
  Mutation rate of ctDNA pre- and post- neoadjuvant chemotherapy and after operation.
Concentration of cfDNA pre- and post- neoadjuvant chemotherapy and after operation. | 2 years
  Concentration of cfDNA pre- and post- neoadjuvant chemotherapy and after operation.
The relationship between tumor response and changes in numbers of CTC pre- and post-neoadjuvant chemotherapy and after operation. | 2 years
  The relationship between tumor response and changes in numbers of CTC pre- and post-neoadjuvant chemotherapy and after operation.
The relationship between tumor response and mutation of ctDNA pre- and post-neoadjuvant chemotherapy and after operation. | 2 years
  The relationship between tumor response and mutation of ctDNA pre- and post-neoadjuvant chemotherapy and after operation.

SECONDARY OUTCOMES:
Disease Free Survival(DFS) | 2 years
  The relationship between CTC, ctDNA and cfDNA and DFS in patients with resectable or locally advanced gastric or gastro-oesophageal junction cancer.
Overall survival(OS) | 2 years
  The relationship between CTC, ctDNA and cfDNA and OS in patients with resectable or locally advanced gastric or gastro-oesophageal junction cancer.
Types of tumor-associated DNA in tumor tissues after operation. | 2 years
  Types of tumor-associated DNA in tumor tissues after operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiuda Zhao, Xining, Qinghai, China